CLINICAL TRIAL: NCT00927433
Title: Development and Implementation of a Structured Educational Programme to Increase Patients Knowledge About Fatigue and to Evaluate the Effect of Increased Knowledge on Cancer Patients Experience of Fatigue
Brief Title: Cancer Patients' Knowledge About Fatigue
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Tone Rustøen, Rikshospitalet HF
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Intervention, cancer fatigue
Record Dates: First submitted 2009-06-23; First posted 2009-06-25 (Estimated); Last update posted 2011-06-30 (Estimated); Status verified 2011-06

CONDITIONS: Cancer; Fatigue
Keywords: Fatigue; Cancer; Radiation therapy; Chemotherapy; Hormones; Surgery; Breast cancer
MeSH Terms: conditions — Neoplasms; Fatigue; Breast Neoplasms | interventions — Standard of Care; Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard care (No Intervention): Patients received standard education about fatigue by clinicians.
  Interventions: Behavioral: Psychoeducational intervention for cancer-related fatigue
- Education arm (Experimental): Patients received education on fatigue management in groups of ten patients over two weeks in three two hour sessions.
  Interventions: Behavioral: Psychoeducational intervention for cancer-related fatigue

INTERVENTIONS:
Behavioral: Psychoeducational intervention for cancer-related fatigue — Patients received education on fatigue management in groups of ten patients over two weeks in three two hour sessions
  Other Names: Standard care; Educational intervention

SUMMARY:
Background: Result from an earlier study I carried out in the late 1990 showed that cancer patients were overall well informed about diagnoses, prognoses, symptoms, treatment, side-effects of treatment e.g. pain, nausea and vomiting and hair loss. Their knowledge about fatigue as a side -effect to cancer and cancer treatment was however different. Patients had minimal knowledge about fatigue and they were not prepared for this side-effect and as a result of this they did not know how to handle fatigue and fatigue was seen as a very frightening experience.

As a result of the findings I wanted to carry out an intervention study, where the aims were to develop an educational programme about fatigue and to evaluate the effect of the programme.

Purpose: The purpose of the project is to develop and describe a structured educational programme. The structured educational programme will serve as the intervention. The purpose is also to evaluate whether or not the structured educational programme increase the cancer patients knowledge about cancer related fatigue and to find out if increased knowledge about cancer related fatigue ease the experience of cancer related fatigue.

Another purpose of the study is to investigate the connection between fatigue and other symptoms and to find out how other symptoms influence the patients experience of fatigue.

The study will consist of 3 stages.

* Development of structured educational programme
* Implementation of structured educational programme
* Evaluation of the effect of the structured educational programme

Materials and methods: The study is a randomised experimental design. An intervention group and a control group, each consisting of 100 Breast Cancer patients (Stadium I or II) receiving chemotherapy or/and radiation therapy after surgery are included in the study. On a NR-scale (0-10) the patients had a fatigue score of 2,5 or more to be included in the study.

The intervention is an educational package of 120 minutes x 3 over three weeks. The intervention is given in groups of 10 patients. Both groups are responding to questionnaires just before the intervention, just after the intervention and three months after finishing the intervention. The educational package consisted of basic knowledge about fatigue, and strategies or techniques for coping with fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Women with breast cancer stage I or II.
* Fatigue score more than 2.5 on a NRS (O-10).
* Give written consent.

Exclusion Criteria:

* Under the age of 10 years,
* Not able to read, write or understand Norwegian.

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2007-10; Primary Completion 2008-03 (Actual); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Level of fatigue | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Tone Rustøen, PhD, Principal Investigator — Oslo University College